CLINICAL TRIAL: NCT05433402
Title: Repurposing the Antipsychotic Drug Chlorpromazine as Adjuvant Therapeutic Agent for Resected Stage III Colon Cancer: A Pilot, Randomized, Open Label, Controlled Study.
Brief Title: Repurposing the Antipsychotic Drug Chlorpromazine as Adjuvant Therapeutic Agent for Resected Stage III Colon Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Organizational safety isues
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Principle Investigator, Sadat City University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Onco-2022-7
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Colon Cancer Stage III
MeSH Terms: conditions — Colonic Neoplasms | interventions — Chlorpromazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Drug: Control
- Chloropromazine (Experimental)
  Interventions: Drug: ChlorproMAZINE 50 MG

INTERVENTIONS:
Drug: ChlorproMAZINE 50 MG — The experimentall group will receive folinic acid, fluorouracil and oxaliplatin (mFOLFOX6) regimen every 14 days for (6-12 cycles) (6 months) (Day 1: 5-FU IV 400 mg/m2, leucovorin IV 400 mg/m2, oxaliplatin IV 85 mg/m2, 5-FU continuous IV infusion (CIVI) 1200 mg/m2/day x 2 days (over 46-48 hours) plus choloropromazine 50 mg daily for 6 months
  Arms: Chloropromazine
Drug: Control — The control group will receive folinic acid, fluorouracil and oxaliplatin (mFOLFOX6) regimen every 14 days for (6-12 cycles) (6 months) (Day 1: 5-FU IV 400 mg/m2, leucovorin IV 400 mg/m2, oxaliplatin IV 85 mg/m2, 5-FU continuous IV infusion (CIVI) 1200 mg/m2/day x 2 days (over 46-48 hours)
  Arms: Control

SUMMARY:
chlorpromazine displays a series of remarkable bio-molecular effects in cancer cells, as inhibition of cell growth, nuclear aberrations, inhibition of the phosphoinositide 3-kinase/mammilian target of rapamycin (PI3K/mTOR) axis, induction of cytotoxic autophagy, inhibition of glutamate and DRD2 receptors. This study will evaluate the addition of chlorpromazine to the first-line therapeutic protocol in colon cancer stage III.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥18 years old.
* Patients with histologically confirmed surgically resected stage III colon cancer
* No rectal cancer
* Stage III disease (any pT, N1-2, M0)
* Patients should have a good performance status according to Eastern Cooperative Oncology Group (ECOG) score (ECOG 0-2).
* Patients with normal organic function as defined for the following criteria:

  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 times the upper normal limit of the local laboratory (LSN-LL);
  * Total serum bilirubin ≤ 2.0 x ULN-LL;
  * Absolute neutrophil count ≥ 1,500 / mm3;
  * Platelet count ≥ 100,000 / mm3;
  * Hemoglobin ≥ 8.0 g / dl;
  * Serum creatinine ≤ 1.5 x ULN-LL
* Patients should undergone curative-intent complete surgical resection
* Patients have at least one month from any major surgery to start of intervention
* Written informed consent before enrollment

Exclusion Criteria:

* Patients with concurrent other malignancy or history of other malignancy treated within the past 3 years (other than non-melanoma skin cancer or in-situ cervical cancer)
* Patients with metastatic disease
* Patients who scheduled to receive any form of further adjuvant cancer therapy (A malignancy currently under active therapy
* Pregnant or breast-feeding patients
* Patients with known hypersensitivity or intolerance to CPZ
* Patients with serious illness or psychiatric condition.
* Patients have current participation in other protocols with experimental drugs.
* Patients with no ability to ingest food orally.
* Patients who have familial adenomatous polyposis, hereditary non-polyposis rectal cancer, or inflammatory bowel disease
* Patients who are taken other chemoprevention drugs (ex. NSAIDs, Aspirin)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | one year
  Disease-free survival as measured by Logrank

SECONDARY OUTCOMES:
Overall survival | one year
  Overall survival as measured by Logrank
Time occurrence of new primary colon cancer and new polyps | one year
  Time occurrence of new primary colon cancer and new polyps as measured by Logrank

OTHER OUTCOMES:
Biological Markers | 6 months
  Blood and serum level of apoptotic and inflammatory markers (Sirtuin 1 (SIRT1) - p53 - TNF-α - Caspase 3)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, University of Sadat city, Madīnat as Sādāt, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF